CLINICAL TRIAL: NCT04541706
Title: SINGLE-ARM STUDY TO EVALUATE THE SAFETY OF LORLATINIB IN ALK INHIBITOR-TREATED UNRESECTABLE ADVANCED AND/OR RECURRENT ALK-POSITIVE NON-SMALL CELL LUNG CANCER PARTICIPANTS IN INDIA
Brief Title: Lorlatinib in ALK Inhibitor Treated Unresectable Advanced/Recurrent ALK-Positive Non Small Cell Lung Cancer Patients in India
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B7461030
Record Dates: First submitted 2020-08-21; First posted 2020-09-09 (Actual); Results first posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-11

CONDITIONS: Advanced Non-Small Cell Lung Cancer
MeSH Terms: interventions — lorlatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lorlatinib (Experimental): The recommended dosage of lorlatinib is 100 mg orally once daily, with or without food, until disease progression, unacceptable toxicity, or participant refusal/lost to follow-up. About 100 participants will be enrolled in this study.
  Interventions: Drug: Lorlatinib

INTERVENTIONS:
Drug: Lorlatinib — Lorlatinib will be supplied for oral administration as 25 mg tablets. The recommended dosage of lorlatinib is 100 mg orally once daily.
  Other Names: LORBRIQUA

SUMMARY:
Lorlatinib is a third-generation, oral, reversible, ATP-competitive, macrocyclic TKI of ALK and ROS1. Lorlatinib was specifically designed to penetrate the CNS and to overcome known secondary resistance mutations in the ALK tyrosine kinase domain.

This is a Phase 4, open-label, multicenter, non-randomized, prospective, single arm study to evaluate the safety and tolerability of lorlatinib in adult participants with unresectable advanced and/or recurrent ALK-positive NSCLC with resistance or intolerance to at least 1 prior ALK inhibitor treatment.

This study is being conducted as a post approval study to fulfill Central Drugs Standard Control Organization (CDSCO) request relating to additional information on use of Lorlatinib in Indian patients.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of histologically or cytologically confirmed diagnosis of unresectable advanced and/or recurrent NSCLC that carries an ALK rearrangement, as detected by an appropriate test.
2. Disease progression or intolerance to 1 previous treatment with ALK TKI. Participants may have also had prior chemotherapy for their advanced and/or recurrent disease.
3. Participants with asymptomatic CNS metastases (including participants controlled with stable or decreasing steroid use within the last 2 weeks prior to study enrollment) will be eligible.
4. Age ≥18 years.
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2.
6. Adequate hematologic and renal function as defined as:

   1. Absolute neutrophil count (ANC) ≥1,000/mm3;
   2. Platelets ≥50,000/mm3;
   3. Hemoglobin ≥8 g/dL;
   4. Estimated creatinine clearance ≥30 mL/min as calculated using the method standard for the institution.
7. Adequate liver function, including:

   1. Total serum bilirubin ≤1.5 × upper limit of normal (ULN);
   2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 × ULN (≤5.0 × ULN in case of liver metastases).
8. Adequate pancreatic function, including:

   1. Serum total amylase ≤1.5 × ULN.*
   2. Serum lipase <1.5 × ULN. *if total amylase >1.5 × ULN, but pancreatic amylase is within the ULN, the participant may be enrolled.
9. Acute effects of any prior therapy resolved to baseline severity or to CTCAE Grade <1 except for AEs that in the Investigator's judgment do not constitute a safety risk for the participant.
10. Systemic anticancer therapy completed within a minimum of 5 half-lives of study enrollment (unless clinically meaningful tumor flare per discretion of the Investigator, in which discussion with the Sponsor is warranted).
11. Evidence of a personally signed and dated informed consent document indicating that the participant (or a legally acceptable representative) has been informed of all pertinent aspects of the study.
12. Willingness and ability to comply with the study scheduled visits, treatment plans, laboratory tests and other procedures.
13. Pregnancy test for females of childbearing potential negative at Screening or female participants who are not of childbearing potential. Male and female participants of childbearing potential and at risk for pregnancy must agree to use a highly effective method of contraception from the time of Screening, throughout the study and for 3 months after the last dose of assigned treatment, 6 months if female participants.

Exclusion Criteria:

1. Radiation therapy (except palliative to relieve bone pain) within 2 weeks of study enrollment. Palliative radiation (<10 fractions) must have been completed at least 48 hours prior to study enrollment. Stereotactic or small field brain irradiation must have completed at least 2 weeks prior to study enrollment. Whole brain radiation must have completed at least 4 weeks prior to study enrollment. Prior irradiation to >25% of the bone marrow.
2. Major surgery within 4 weeks prior to enrollment. Minor surgical procedures (eg, port insertion) are not excluded, but sufficient time should have passed for adequate wound healing.
3. Known prior or suspected severe hypersensitivity to study drug or any component in its formulation.
4. Active and clinically significant bacterial, fungal, or viral infection.
5. Clinically significant vascular (both arterial and venous) and non-vascular cardiac conditions (active or within 3 months prior to enrollment), which may include, but are not limited to:

   1. Arterial disease such as cerebral vascular accident/stroke (including transient ischemic attack [TIA]), myocardial infarction, unstable angina;
   2. Venous diseases such as cerebral venous thrombosis, symptomatic pulmonary embolism;
   3. Non-vascular cardiac disease such as congestive heart failure (New York Heart Association Classification Class ≥II), second degree or third degree atrioventricular (AV) block (unless paced) or any AV block with PR interval >220 msec; or ongoing cardiac dysrhythmias of NCI CTCAE Grade ≥2, uncontrolled atrial fibrillation of any grade, bradycardia defined as <50 beats per minute (bpm) (unless participant is otherwise healthy such as long distance runners, etc.), machine read ECG with QT interval corrected for heart rate (QTc) >470 msec, or congenital long QT syndrome.
6. History or known presence of interstitial fibrosis, interstitial lung disease (ILD), pneumonitis, hypersensitivity pneumonitis, interstitial pneumonia, obliterative bronchiolitis, and pulmonary fibrosis.
7. Other severe acute or chronic medical or psychiatric condition, including recent (within the past year) or active suicidal ideation or behavior, or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the participant inappropriate for enrollment in this study.
8. Evidence of active malignancy (other than current NSCLC, non-melanoma skin cancer, in situ cervical cancer, papillary thyroid cancer, ductal carcinoma in situ [DCIS] of the breast or localized and presumed cured prostate cancer) within the last 3 years prior to enrollment.
9. Concurrent use of any of the following food or drugs (consult the Sponsor if in doubt whether a food or a drug falls into any of the categories described below) within 12 days prior to the first dose of lorlatinib:

   1. Known strong cytochrome (CYP)3A inducers (eg, carbamazepine, enzalutamide, mitotane, rifampin, St. John's Wort).
   2. Known strong CYP3A inhibitors (eg, grapefruit juice or grapefruit/grapefruit related citrus fruits [eg, Seville oranges, pomelos], boceprevir, cobicistat, clarithromycin, conivaptan, diltiazem, idelalisib, indinavir, itraconazole, ketoconazole, lopinavir, nelfinavir, paritaprevir, posaconazole, ritonavir alone and with elvitegravir or indinavir or lopinavir or paritaprevir or ombitasvir or dasabuvir or saquinavir or tipranavir, telaprevir and voriconazole). The topical use of these medications (if applicable), such as 2% ketoconazole cream, is allowed.
   3. Known CYP3A substrates with narrow therapeutic index, such as pimozide, quinidine, tacrolimus, cyclosporine, sirolimus, alfentanil, fentanyl (including transdermal patch) or ergot alkaloids (ergotamine, dihydroergotamine).
   4. Known permeability glycoprotein (P-gp) substrates with a narrow therapeutic index (eg, digoxin).
10. Participants who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the Investigator, or participants who are Pfizer employees directly involved in the conduct of the study.
11. Participation in other studies involving investigational drug(s) (Phases 1-4) during study participation.
12. Breastfeeding female participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- India (12):
  - The Gujarat Cancer and Research Institute, Ahmedabad, Gujarat
  - Hemato Oncology Clinic Ahmedabad Pvt. Ltd, Ahmedabad, Gujarat
  - Artemis hospital, Gurugram, Haryana
  - National Cancer Institute, Nagpur, Maharashtra
  - Apex Wellness Hospital, Nashik, Maharashtra
  - Grant Medical Foundation, Ruby Hall Clinic, Pune, Maharashtra
  - Sahyadri Clinical Research and Development Center, Pune, Maharashtra
  - Sahyadri Super Speciality Hospital, Pune, Maharashtra
  - Bhaktivedanta Hospital and Research Institute, Thane, Maharashtra
  - Rajiv Gandhi Cancer Institute And Research Centre, New Delhi, National Capital Territory of Delhi
  - Yashoda Hospital, Hyderabad, Telangana State
  - Tata Medical Center, Kolkata, West Bengal

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7461030

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 111 participants were screened, 10 participants had screen failure and 1 participant died before enrollment, 100 participants were enrolled and received treatment.
Groups:
- Lorlatinib 100 mg QD: Participants received lorlatinib 100 mg (4 x 25 mg tablets swallowed whole) orally once daily (QD) until disease progression, unacceptable toxicity, or participant refusal/lost to follow-up.
Period: Overall Study
Arm/Group | Lorlatinib 100 mg QD
Started | 100
Completed | 55
Not Completed | 45
Not completed — Withdrawal by Subject | 3
Not completed — Progressive disease | 33
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 2
Not completed — Death | 5
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all participants enrolled and treated in the study.
Arm/Group | Lorlatinib 100 mg QD
Number analyzed (Participants) | 100
Age, Continuous [Median (Full Range); unit: Years] | 49.0 [24.0 to 77.0]
Age, Customized [Number; unit: Participants]
  <18 years | 0
  18-44 years | 38
  45-64 years | 47
  >=65 years | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 60
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 100
  American India or Alaska Native | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a product or medical device; the event did not necessarily need to have a causal relationship with the treatment or usage. A TEAE was defined as an event that emerged during treatment, having been absent pretreatment, or worsened relative to the pretreatment state. If the investigator did not know whether or not the investigational product caused the event, then the event would be handled as "related to investigational product" for reporting purposes, as defined by the sponsor. If the investigator's causality assessment was "unknown but not related to investigational product," this was clearly documented on study records.
Time Frame: From Day 1 up to 35 days post last dosing date or the date of initiation of a new anticancer therapy (up to 1.9 years)
Population: The safety analysis population included participants who received at least 1 dose of lorlatinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib 100 mg QD
Number analyzed (Participants) | 100
Participants
  All-causality TEAEs | 94
  Treatment-related TEAEs | 89

2. Secondary Outcome: Confirmed Objective Responses Rate (ORR) Based on Investigator Assessment
Description: ORR was defined as the percentage of participants with best overall response as confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. ORR was provided along with the corresponding 95% confidence interval (CI) based on Wilson's Score Method. CR was defined as the disappearance of all target lesions. PR was defined as at least a 30% decrease in the sum of the target lesions.
Time Frame: Assessed at least 1 year from first dose or until progression of disease, death or received subsequent anti-cancer therapy, whichever came first up to a maximum of 2 years.
Population: The analysis population included participants who received at least 1 dose of lorlatinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lorlatinib 100 mg QD
Number analyzed (Participants) | 100
Percentage of participants | 41 [31.9 to 50.8]

3. Secondary Outcome: Confirmed Intracranial Objective Response Rate (IC-ORR) Based on Investigator Assessment
Description: IC-ORR was defined as the percentage of participants with intracranial response (ie, best overall intracranial response as confirmed CR or confirmed PR considering only intracranial lesions) relative to participants with central nervous system (CNS) metastases at study entry. IC-ORR was provided along with the corresponding 95% CI based on Wilson's Score Method. CR was defined as the disappearance of all target lesions. PR was defined as at least a 30% decrease in the sum of the target lesions.
Time Frame: as for outcome 2
Population: The analysis population included participants any intracranial lesions.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lorlatinib 100 mg QD
Number analyzed (Participants) | 56
Percentage of participants | 35.7 [24.5 to 48.8]

4. Secondary Outcome: Duration of Response (DoR)
Description: DoR was defined as the time from the first documentation of objective tumor response (confirmed CR or confirmed PR) to the first documentation of disease progression or death due to any cause, whichever occurred first. For participants whose responses proceed from PR to CR, the onset of PR was taken as the onset of response. CR was defined as the disappearance of all target lesions. PR was defined as at least a 30% decrease in the sum of the target lesions.
Time Frame: as for outcome 2
Population: The analysis population included participants with confirmed objective response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lorlatinib 100 mg QD
Number analyzed (Participants) | 41
Months | NA [NA to NA] — The median DoR was not reached. The survival curve for the DoR did not reach 50% so the median and 95%CI could not be calculated. This was due to having participants who had the highest survival times and had yet to experience the event/disease progression.

5. Secondary Outcome: Intracranial Duration of Response (IC-DoR)
Description: IC-DoR was defined as the time from the first documentation of an intracranial objective response (confirmed CR or confirmed PR) to the first documentation of disease progression or death due to any cause, whichever occurred first in the subgroup of participants with brain metastasis at baseline. CR was defined as the disappearance of all target lesions. PR was defined as at least a 30% decrease in the sum of the target lesions.
Time Frame: as for outcome 2
Population: The analysis population included participants with CNS metastases at baseline and confirmed objective response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lorlatinib 100 mg QD
Number analyzed (Participants) | 20
Months | NA [11.1 to NA] — The median DoR was not reached. The survival curve for the DoR did not reach 50% so the median and 95%CI could not be calculated. This was due to having participants who had the highest survival times and had yet to experience the event/disease progression.

ADVERSE EVENTS:
Time Frame: From Day 1 up to 35 days post last dosing date or the date of initiation of a new anticancer therapy (up to 1.9 years)
Description: The same event may appear as both an AE and a serious AE (SAE). An event may be categorized as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Arm/Group | Lorlatinib 100 mg QD
All-Cause Mortality (participants affected / at risk) | 8/100
Serious Adverse Events (participants affected / at risk) | 22/100
Other Adverse Events (participants affected / at risk) | 89/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lorlatinib 100 mg QD (N=100)
Cardiac arrest (Cardiac disorders) | 1
Cardiac tamponade (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Sudden death (General disorders) | 1
COVID-19 (Infections and infestations) | 4
COVID-19 pneumonia (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Pneumonia aspiration (Infections and infestations) | 1
Suspected COVID-19 (Infections and infestations) | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Altered state of consciousness (Nervous system disorders) | 1
Cognitive disorder (Nervous system disorders) | 1
Hypersomnia (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Acute psychosis (Psychiatric disorders) | 1
Mania (Psychiatric disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lorlatinib 100 mg QD (N=100)
Anaemia (Blood and lymphatic system disorders) | 26
Oedema (General disorders) | 7
Oedema peripheral (General disorders) | 29
Peripheral swelling (General disorders) | 6
COVID-19 (Infections and infestations) | 6
Weight increased (Investigations) | 39
Dyslipidaemia (Metabolism and nutrition disorders) | 7
Hypercholesterolaemia (Metabolism and nutrition disorders) | 57
Hyperglycaemia (Metabolism and nutrition disorders) | 16
Hyperlipidaemia (Metabolism and nutrition disorders) | 20
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 58
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8
Hypertension (Vascular disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-03-30): https://cdn.clinicaltrials.gov/large-docs/06/NCT04541706/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-03): https://cdn.clinicaltrials.gov/large-docs/06/NCT04541706/SAP_001.pdf